CLINICAL TRIAL: NCT01125761
Title: Efficacy and Safety of the Association of Dexamethasone 0.5 mg + Clemastine Fumarate 1 mg When Compared to Dexamethasone 0.5 mg in Patients With Allergic Dermatitis
Brief Title: Efficacy and Safety of the Association Drugs in Patients With Allergic Dermatitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DECEMS21209
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Dermatitis
Keywords: Allergic dermatitis
MeSH Terms: conditions — Dermatitis; Dermatitis, Atopic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone 0.5 mg and 1.0 mg clemastine cream (Experimental)
  Interventions: Drug: dexamethasone 0.5 mg and 1.0 mg clemastine cream
- dexamethasone 0,5 mg cream (Active Comparator)
  Interventions: Drug: Dexamethasone 0,5 mg cream

INTERVENTIONS:
Drug: dexamethasone 0.5 mg and 1.0 mg clemastine cream — The treatment should be administered every 12 hours so that a thin layer is applied on the lesions, for 14 days.
  Arms: dexamethasone 0.5 mg and 1.0 mg clemastine cream
Drug: Dexamethasone 0,5 mg cream — The treatment should be administered every 12 hours so that a thin layer is applied on the lesions, for 14 days.
  Arms: dexamethasone 0,5 mg cream

SUMMARY:
Considering the pathogenesis of several allergic skin diseases to be investigated in this study as well as the pharmacodynamic mechanisms of the association of dexamethasone and clemastine fumarate, it is believed that the components of topical medication may act synergistically in the reduction of signs and symptoms of the diseases in question. Therefore it is expected that the association promotes results significantly superior to dexamethasone alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients who sign the Deed of Consent (IC) in two ways, by his own free will, agreeing with all study procedures;

  * Patients older than 18 years, any ethnicity, class or social group, regardless of sex;
  * Patients with pictures of dermatoses acute, subacute or chronic, of inflammatory origin and / or allergic, to which it is recommended the use of drugs under investigation topically, such as:
* atopic dermatitis,
* prurigo,
* primary contact dermatitis or allergic
* urticaria,
* pharmacodermic,
* allergic vasculitis,
* dyshidrosis,

Exclusion Criteria:

* Patients being treated with antibiotics;
* Participation in clinical trials in the 12 months preceding the survey;
* Current treatment with immunosuppressants (eg, cyclosporine or methotrexate);
* Current treatment with phototherapy (UVA, UVB, PUVA and lasers);
* Use of systemic corticosteroids at inclusion visit or within 15 days prior to inclusion;
* Topical treatments at the site of acne in the 15 days preceding the visit of inclusion;
* Presence of any skin condition in areas affected by acne that hamper the evolutionary analysis of the lesion;
* Presence of secondary infections at the site of treatment, diagnosed clinically;
* Presence of other eczematous picture, such as nummular eczema, neurodermatitis, seborrheic dermatitis, psoriasis, scabies, and Buckley's syndrome Wiskott-Aldrich;
* Pregnant or lactating women;
* Chronic alcoholism;
* Patients with a history of hypersensitivity to any component of the formulas of the products under investigation;
* Any finding of clinical observation (clinical history or physical examination) that is interpreted by the physician investigator as a risk to the patient's participation in the study;
* Allergic Dermatosis of moderate or severe that, according to the investigator, is not justified topical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11

PRIMARY OUTCOMES:
Through clinical examinations, evaluating the efficacy of the cream composed by 0.5 mg dexamethasone and clemastine 1mg compared with the cream of 0.5 mg dexamethasone in improving the signs and symptoms associated with allergic dermatitis. | 14 days

SECONDARY OUTCOMES:
Improvement of the erythema associated with allergic dermatitis. | 14 days
Improvement of the edema associated with allergic dermatitis. | 14 days
Improvement of the extension of lesion associated with allergic dermatitis. | 14 days
Evaluate, through clinical examinations, the effectiveness of the drug association in reducing excoriation associated with allergic dermatitis. | 14 days
Evaluate, through clinical examinations, the effectiveness of the drug association in reducing exudation associated with allergic dermatitis. | 14 dyas
Evaluate, through clinical examinations, the effectiveness of the drug association in reducing of scabbing associated with allergic dermatitis. | 14 days
Evaluate, through clinical examinations, the effectiveness of the drug association in reducing of lichenification associated with allergic dermatitis. | 14 days
Evaluate the safety of the formulations in relation to the occurrence, type, frequency and intensity of adverse events during treatment. | 14 days

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - LAL Clinica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo
  - LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo